CLINICAL TRIAL: NCT02822482
Title: Phase ib/II Trial of Copanlisib, a Selective PI3K Inhibitor, in Combination With Cetuximab in Patients With Recurrent and/or Metastatic (R/M) Head and Neck Squamous Cell Carcinoma (HNSCC) Harboring a PI3KCA Mutation/Amplification and/or a PTEN Loss.
Brief Title: Copanlisib in Association With Cetuximab in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinomas Harboring a PI3KCA Mutation/Amplification and/or a PTEN Loss
Acronym: COPAN-ORL06
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: futilty of the treatment
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0130/1507; 2015-004340-19 (EudraCT Number)
Record Dates: First submitted 2016-06-16; First posted 2016-07-04 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — copanlisib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copanlisib + Cetuximab (Experimental): All patients will be treated by Copanlisib in association with Cetuximab.
  Interventions: Drug: Copanlisib; Drug: Cetuximab

INTERVENTIONS:
Drug: Copanlisib — Copanlisib will be given at Day 1, Day 8 and Day 15 (1 cycle = 28 days), administered intravenously over 60 minutes, in association with Cetuximab.
  Other Names: BAY 80-6946
Drug: Cetuximab — Cetuximab will be given weekly at Day 1, Day 8, Day 15 and Day 22 (1 cycle = 28 days), administered intravenously over 120 minutes (Cycle 1 Day 1) or 60 minutes (subsequent infusions), in association with Copanlisib.
  Other Names: Erbitux

SUMMARY:
The study consists of two distinct and sequential parts:

* A Phase Ib aimed at determining the MTD (Maximum Tolerated Dose) of the combination (copanlisib/cetuximab) and the RP2D
* A Phase II aimed at evaluating the efficacy of the combination at the RP2D (Recommended Phase 2 Dose)

All patients will be treated with the Copanlisib, a selective PI3KCA inhibitor, in association with Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with R/M HNSCC (oropharynx, oral cavity, hypopharynx and larynx), histologically or cytologically confirmed, not amenable to curative treatment with surgery and/or chemotherapy and/or radiotherapy (Stage III/IV)
2. Adult men and women ≥ 18 years
3. Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
4. Patients with tumor harboring a PI3K mutation/amplification and/or a PTEN loss
5. Patients with a radiologic documented progression or relapse after cetuximab therapy (patients could have either received combination platinum doublet with cetuximab or cetuximab after platinum doublet)
6. Patients with prior platinum based therapy, unless contraindicated
7. Patients with at least one measurable lesion assessed by Magnetic Resonance Imaging (MRI) or a computerized tomography scanner (CT-scan) according to RECIST v1.1. Patients must have clinically and/or radiographically documented measurable disease. At least one site of disease must be unidimensionally measurable as follows

   * CT-scan, physical exam ≥ 10 mm
   * Lymph node short axis ≥ 15 mm Tumor measurements must be performed within 28 days prior to starting study drug
8. Women of childbearing potential and men must agree to use adequate contraception when sexually active. This applies since signing of the informed consent form and up to 12 months (for women of child bearing potential) and 6 months (for fertile men) after the last study drug administration (Copanlisib). Highly effective contraception methods are detailed in section 7.2
9. Women of childbearing age or sexually active female patients with reproductive potential must have a negative pregnancy test (serum or urine within the 7 days prior to starting study drug)
10. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
11. Patients with social insurance coverage
12. Glomerular filtration rate (GFR) ≥ 40 mL/min/1.73 m² according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula (within 7 days prior to starting study drug). If not on target, this evaluation may be repeated once after at least 24 hours either according to the MDRD abbreviated formula or by 24 hour sampling. If the later result is within acceptable range, it may be used to fulfill the inclusion criteria instead

Exclusion Criteria:

1. Patients previously treated with PI3K and/or mTOR inhibitors
2. Patients with anticancer therapy (radiotherapy, immunotherapy, chemotherapy, etc.) within 28 days or investigational treatment within 28 days prior to the initiation of study drug treatment, unless evidence of progression since last treatment
3. Patients currently using other approved or investigational anti-neoplasic agent
4. Patients with uncontrolled arterial hypertension despite optimal medical management, Congestive heart failure > New York Heart Association (NYHA) class 2, Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of test drug No active cardiac disease including any of the following: left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO) and QTc > 470 ms on screening ECG
5. Patients with uncontrolled diabetes mellitus (patients with controlled Type I or II diabetes mellitus will be eligible but only into the phase II of the study and only if fasting HbA1c ≤ 8.5% at screening)
6. Patients with a history of Human Immunodeficiency Virus (HIV) Hepatitis B (HBV) or hepatitis C (HCV) infection. All patients must be screened for HIV, HBV and HCV up to 28 days prior to first dosing using the routine virus laboratorial panel. Patients who are positive for HBs Ag or HBc Ab will be eligible if they are negative for HBV-DNA. Patients who are positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA
7. Patients with active uncontrolled or symptomatic central nervous system (CNS) metastases. Patients are eligible if their disease is controlled at least 30 days on corticosteroids prior to starting study drug
8. Patients with major surgery within 28 days, or open biopsy within 7 days, prior to starting study drug. Patients must have recovered from major side effects of the surgery
9. Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible. Copanlisib is primarily metabolized by CYP3A4. Therefore concomitant use of strong inhibitors of CyP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and inducers of CYP3A (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, st. John's Wort) are not permitted from Day -14 of Cycle 1 until the Safety follow up visit
10. Patients with altered hematopoietic or organ function, as indicated by the following criteria (assessed within 7 days prior the first dosing):

    * Absolute granulocytes < 1.0 x 10⁹/L
    * Platelets < 75 x 10⁹/L
    * ALAT/ASAT > 2.5 x ULN in the absence of or > 5 x ULN in the presence of liver metastases
    * Bilirubin > 1.5 x ULN (except Gilbert Syndrome: < 3.0 mg/dL)
    * Creatinine clearance < 60 mL/min (measured or calculated by Cockcroft and Gault formula) or serum creatinine > 1.0 x ULN
    * Lipase > 1.5 x ULN
    * INR and PTT > 1.5 x ULN
11. Patients with a history of hypersensitivity to other monoclonal antibodies or to the active or inactive excipients of study drug
12. Known drug or alcohol abuse
13. Known or underlying medical condition that, in the investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or adverse events
14. History of uncontrolled seizures, seizure disorder requiring medication, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake
15. Unwillingness to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study
16. Individuals deprived of liberty or placed under the authority of a tutor
17. Previous or concurrent history of malignancies within 5 years prior to study treatment except for curatively treated:

    * Cervical carcinoma in situ
    * Non-melanoma skin cancer
    * Superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
    * Localized prostate cancer
18. Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication
19. Proteinuria of ≥ CTCAE Grade 3 as assessed by a 24h protein quantification or estimated by urine protein-creatinine ratio > 3.5 on a random urine sample
20. History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
21. Concurrent diagnosis of pheochromocytoma
22. Pregnant or breast-feeding patients. Women of childbearing potential must have a serum pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment
23. Unresolved toxicity higher than CTCAE Grade 1 attributed to any prior therapy/procedure, excluding alopecia
24. Ongoing immunosuppressive therapy
25. Blood or platelets transfusion less than 7 days before starting treatment
26. Myeloid growth factors within 14 days prior to treatment
27. Systemic continuous corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not allowed. Previous corticosteroid therapy must be stopped or reduced to the allowed dose 7 days before performing the screening CT scan/MRI, whichever is performed first, and again prior to the first study drug administration. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose after the patient has signed the IC. Patients may be using topical or inhaled corticosteroids
28. History of having received an allogeneic bone marrow or organ transplant
29. Anti-arrhythmic therapy (beta blockers or digoxin are permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Phase Ib (dose escalation phase): to determine the Maximal Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of Copanlisib in association with Cetuximab | 1 month
  Determination of the MTD will be based on the occurence of Dose Limiting Toxicities during Cycle 1.
Phase II (expansion phase) : to assess the efficacy of the combination (Copanlisib + Cetuximab) at the RP2D. | 16 weeks
  Efficacy of the combination will be assessed through Progression Free Survival at week 16.

SECONDARY OUTCOMES:
Efficacy of the combination | Through the study completion with an average of 10 months
  Objective Response Rate (ORR) using RECIST 1.1 criteria
Efficacy of the combination | Through the study completion with an average of 10 months
  Overall Survival (OS)
Adverse Events (NCI CTCAE v4.0) | Up to 15 cycles
  All Adverse Events (NCI CTCAE v4.0), related or not related to Copanlisib or Cetuximab, will be collected in the Case Report Form in order to picture the safety profile of the association.
Copanlisib Maximum Plasma Concentration [Cmax] | First Month (at Day 1 and Day 15)
  For patients enrolled in the phase Ib (dose escalation phase) pharmacokinetic samples (blood) will be collected at Cycle 1 Day 1 and Cycle 1 Day 15. There will be 5 samples per day: pre-infusion, end of infusion, 2 hours, 8 hours and 24 hours after the start of Copanlisib infusion.
Area Under the Curve [AUC] for Copanlisib pharmacokinetic | First Month (at Day 1 and Day 15)
  For patients enrolled in the phase Ib (dose escalation phase) pharmacokinetic samples (blood) will be collected at Cycle 1 Day 1 and Cycle 1 Day 15. There will be 5 samples per day: pre-infusion, end of infusion, 2 hours, 8 hours and 24 hours after the start of Copanlisib infusion.
Mutational profile of circulating tumoral DNA (ctDNA) | through the study duration: baseline, C1D1, C1D15, 8 weeks, disease progression
  For patients enrolled in the phase II (dose escalation phase) blood samples will be collected at baseline, C1D1, C1D15, 8 weeks, Disease progression or end of treatment whichever comes first.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Lorraine, Nancy
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Marret G, Isambert N, Rezai K, Gal J, Saada-Bouzid E, Rolland F, Chausson M, Borcoman E, Alt M, Klijanienko J, Vansteene D, Guigay J, Kamal M, Bieche I, Le Tourneau C; UNICANCER Head, Neck Group. Phase I trial of copanlisib, a selective PI3K inhibitor, in combination with cetuximab in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Invest New Drugs. 2021 Dec;39(6):1641-1648. doi: 10.1007/s10637-021-01152-z. Epub 2021 Jul 28. PMID 34322775